CLINICAL TRIAL: NCT05230472
Title: Effect of Statin Therapy on Mortality in Patients With Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanan Mahmoud Farag Awad, hananfarag@med.asu.edu.eg, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EMASU M D 219 /2020
Record Dates: First submitted 2022-01-21; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: VAP - Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated to simvastatin (60 mg) or control given via a nasogastric tube or orally from study inclusion to ICU discharge, death, or day 28, whichever occurred first. Simvastatin or control were started on the same day as antibiotic therapy for suspected VAP. The simvastatin dosage was halved in patients with renal failure (creatinine clearance <30 mL/min). A computer-generated random- number table was prepared by statisticians to assign patients in blocks of 4 to receive either simvastatin or control.
  Block size was unknown to the investigators, who was enrolled the patients and then called the statistics department to obtain the randomization and treatment numbers after checking the inclusion and non-inclusion criteria.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Block size was unknown to the investigators, who was enrolled the patients and then called the statistics department to obtain the randomization and treatment numbers after checking the inclusion and non-inclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- simvastatin group (Active Comparator): 68 patients who had a ventilator associated pneumonia received simvastatin
  Interventions: Drug: Simvastatin
- control group (No Intervention): 68 patients who had a ventilator associated pneumonia not received simvastatin

INTERVENTIONS:
Drug: Simvastatin — simvastatin 60 mg tab
  Arms: simvastatin group

SUMMARY:
Statins with their powerful anti-inflammatory, immunomodulatory, and antioxidant properties make them candidate members to be used in the management of sepsis and different types of infections including pneumonia.

This study aims to determine whether adjunctive statin therapy decreased day- 28 mortality among ICU patients with ventilator-associated pneumonia (VAP) & number of ventilator-free days (after successful weaning) between day 1 and both day 28.

DETAILED DESCRIPTION:
This prospective randomized control-controlled triple blind study was conducted on above 18 years who had received mechanical ventilation in the ICU for at least 2 days.

All included cases were subjected to:

* Demographic data,
* Physiological variables
* Simplified Acute Physiology Score II at admission and radiologic score (Weinberg et al., 1984).
* Antibiotics used, and relevant diagnostic and therapeutic interventions in the ICU.
* The Sequential Organ Failure Assessment (SOFA) score and Clinical Pulmonary Infection Score (CPIS) were calculated on the day of enrolment (day 1) and then on days 3, 7, and 14. Patients were monitored daily for evidence of infection.
* The duration of mechanical ventilation, length of ICU stay, and length of hospital stay were recorded.
* The occurrence of myocardial ischemia or infarction was assessed until day 28. Serum levels of creatine kinase, ALT, and AST were measured.

Patients were randomly allocated to simvastatin (60 mg) or control given via a nasogastric tube or orally from study inclusion to ICU discharge, death, or day 28, whichever occurred first. Simvastatin or control were started on the same day as antibiotic therapy for suspected VAP. The simvastatin dosage was halved in patients with renal failure (creatinine clearance <30 mL/min). A computer-generated random- number table was prepared by statisticians to assign patients in blocks of 4 to receive either simvastatin or control.

Block size was unknown to the investigators, who was enrolled the patients and then called the statistics department to obtain the randomization and treatment numbers after checking the inclusion and non-inclusion criteria Outcome The primary outcome was the day-28 mortality rate. Secondary outcomes were ICU mortality rates; number of days outside the ICU between day 1 and day 28; and number of ventilator-free days (after successful weaning) between day 1 and both day 28.

Successful weaning was defined as spontaneous breathing for at least 48 hours after disconnection of the ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suspected to had VAP defined as a modified Clinical Pulmonary Infection Score (CPIS) of at least 5 and if they underwent quantitative bacteriological cultures of bronchoalveolar lavage (BAL) fluid, a protected telescopic catheter (PTC), or an endotracheal aspirate. The modified CPIS is based on body temperature, blood leukocyte count, amount and appearance of tracheal secretions, ratio of partial pressure of oxygen (PaO2) to fraction of inspired oxygen, acute respiratory distress syndrome (ARDS), and infiltrates on chest radiography. The total can range from 1 to 10 points (Luna et al., 2003).
* Patients were included only for the first episode of suspected VAP.

Exclusion Criteria:

* o Statin therapy at intubation

  * Previous VAP episode during the same hospitalization
  * Known pregnancy
  * Immunodepression with bone marrow aplasia
  * Imminent death (Simplified Acute Physiology Score II of 75 or greater, calculated over the last 6 hours)
  * Treatment limitation decisions
  * Nothing-by-mouth order and no nasogastric tube, continuous gastric aspiration
  * Known chronic intestinal malabsorption
  * Known simvastatin hypersensitivity
  * Acute hepatic failure
  * Use of CYP3A4 inhibitors or cyclosporine
  * Creatine kinase level greater than 5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels greater than 3 times the upper limit of normal

Ages: 29 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the day-28 mortality rate. | 28 day
  asses effect of statin on mortality in ventilator associated pneumonia patient

SECONDARY OUTCOMES:
ICU mortality rates | between day 1 and day 28
  rate of mortality of patients with ventilator associated pneumonia between simvastatin group and control group in intensive care unit
number of days outside the ICU between day 1 and day 28 | between day 1 and day 28
  the number of days patients who have improved spent outside the icu between day 1 and day 28
number of ventilator-free days (after successful weaning) between day 1 and both day 28. | between day 1 and day 28
  number of days patient of the two group spent without ventilator in the intensive care unit between day 1 and day 28 after successful weaning. Successful weaning was defined as spontaneous breathing for at least 48 hours after disconnection of the ventilator.

CONTACTS AND LOCATIONS:
Overall Officials: YOUSEF FAWZY, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No